CLINICAL TRIAL: NCT01513850
Title: A 52-week, Multi-center, Open Label, Single Arm, Phase 3 Study to Evaluate the Efficacy and Safety of Hepabulin IV in HBsAg Positive Liver Transplantation Recipients
Brief Title: A Confirmatory Study of Hepabulin IV in HBsAg Positive Liver Transplantation Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hepabulin IV_LT_lll_2011
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis B
Keywords: Liver Transplantation; HBV; HBV Recurrence; HBsAg Positive
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepabulin IV (Experimental)
  Interventions: Drug: Hepabulin IV

INTERVENTIONS:
Drug: Hepabulin IV — I.V.

SUMMARY:
The purpose of this study is to Evaluate the efficacy and safety of Hepabulin IV (HBIG, a study drug) after liver transplantation.

DETAILED DESCRIPTION:
A 52-week, Multi-center, Open label, Single arm, Phase 3 Study to Evaluate the Efficacy and Safety of Hepabulin IV in HBsAg positive Liver Transplantation recipients

ELIGIBILITY:
Inclusion Criteria:

* HBsAg Positive candidate for HBV-related liver transplant
* Primary, single organ recipients
* written informed consent

Exclusion Criteria:

* acute renal failure, Serum creatinin >1.5*ULN
* severe cardiac disease or other significant disease
* HAV, HCV or HIV positive
* Immunoglobulin A deficiency.
* History of hypersensitivity to Human Immunoglobulin.
* History of cancer within 5 years. (without HCC)
* History of alcohol or/and drug abuse.
* History organ transplantation.
* Within 30 days, participation in another clinical trial and use of an investigational product.
* Subject suffer from any acute or chronic medical, surgical or psychiatric condition or laboratory abnormality that, may increase the risk associated with the study participation or investigational product administration, or may interfere with the interpretation of study result.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
HBV(HBsAg) recurrence | 52 weeks

SECONDARY OUTCOMES:
Time to recurrence | 52 weeks
Survival | 52 weeks
viral Marker of HBV | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong Goo Kim, MD, PhD, Study Chair — St.Mary's Hospital, Catholic University Medical college
Locations (1):
- SKChemicals, Seongnam, Gyunggi-do, South Korea